CLINICAL TRIAL: NCT03093636
Title: Efficacy of inControl Advice: A Decision Support System (DSS) for Diabetes
Acronym: DSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: TypeZero Technologies (Industry); Novo Nordisk A/S (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19634; DP3DK101055 (NIH); U1111-1191-3911 (Other: Universal Trial Number)
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus (T1DM); Continuous Glucose Monitor (CGM); Multiple Daily Injections (MDI); Insulin Pen; inControl Advice; Decision Support System (DSS)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Continuous Glucose Monitor (CGM)+Decision Support System (DSS) (Experimental): Continuous Glucose Monitor (CGM)+Decision Support System (DSS) study participants will use the inControl Advice App, study insulin, and study CGM at home for 12 weeks.
  Interventions: Device: Continuous Glucose Monitor (CGM)+Decision Support System (DSS)
- Continuous Glucose Monitor (CGM) alone (Placebo Comparator): Continuous Glucose Monitor (CGM) alone study participants will use study insulin and the study CGM alone at home for 12 weeks.
  Interventions: Other: Continuous Glucose Monitor (CGM) alone

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM)+Decision Support System (DSS) — Continuous Glucose Monitor (CGM)+Decision Support System (DSS) study participants will use the inControl Advice App and a study CGM at home for 12 weeks. The DSS contains a "smart" bolus advisor that adjusts the size of the correction insulin boluses based on short-term blood glucose predictions. It is able to complete this function by evaluating CGM values, insulin usage and carbohydrate intake record. It also contains an exercise advisor, a bedtime advisor, hypoglycemia risk and long-term tracker of HbA1c. Subjects will use study basal and bolus insulin during the study.
  Arms: Continuous Glucose Monitor (CGM)+Decision Support System (DSS)
Other: Continuous Glucose Monitor (CGM) alone — Continuous Glucose Monitor (CGM) alone study participants will use a study CGM at home for 12 weeks. Subjects will use study basal and bolus insulin during the study.
  Arms: Continuous Glucose Monitor (CGM) alone

SUMMARY:
The purpose of this study is to reduce the frequency of hypoglycemia and severe hypoglycemic events in subjects who use insulin pens to treat their Type 1 Diabetes Mellitus (T1DM). Hypoglycemia is the number one fear of many individuals and families with someone who has type 1 diabetes, and this fear often prevents optimal glycemic control. It is expected that this protocol will yield increased knowledge about using a decision support system to help control the glucose level.

DETAILED DESCRIPTION:
This study is a 12-week parallel group multi-center randomized trial designed to compare CGM+DSS with CGM alone. The DSS to be implemented contains a "smart" bolus advisor that adjusts the size of correction insulin boluses based on short term blood glucose predictions. It is able to complete this function by evaluating CGM values, insulin usage and carbohydrate intake record. It also contains an exercise advisor, a bedtime advisor, hypoglycemia risk and long-term tracker of HbA1c.

inControl-Advice, a smart-phone based medical software platform, is designed to provide advice to users. It receives data from an insulin pen and then adjustments the insulin delivery every 5 minutes. The system provides a series of real-time alerts and on-demand advice, for both dosing of insulin and ingestion of carbohydrates, based on data collected from T1DM patients (i.e. carbohydrate consumption, insulin injected, CGM) and inConrol Cloud analytics.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide informed consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year
3. Using basal and meal insulin (NovoLog® [insulin aspart], Humalog® [insulin lispro] or Apidra® [insulin glulisine]) for Intensive Insulin Therapy including carbohydrate counting and use of pre-defined parameters for glucose goal, carbohydrate ratio, and insulin sensitivity factor for at least 1 month.

   a. Acceptable basal insulin regimens include: i. Lantus® (insulin glargine) 100U/mL once or twice daily ii. Levemir® (insulin detemir) 100U/mL once or twice daily iii. Tresiba® (insulin degludec) 100U/mL once daily
4. Age ≥15.0 years old
5. Willingness to use the study basal insulin (Tresiba® [insulin degludec]) and meal insulin (NovoLog® [insulin aspart]) for the duration of the study.
6. Willingness to use the home or DSS-optimized carbohydrate counting parameters for all meal dosing and enter the information into the inControl APP (for CGM+DSS group).
7. For females, not currently known to be pregnant
8. If female and sexually active, must agree to use a highly effective form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study. Also, subjects who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
9. Ability to access the Internet to provide data to the clinical team or to travel to the research center so that the study equipment can be downloaded.
10. Ability to have 3G or Wi-Fi to be able to use the DSS smart bolus calculator and advice given (i.e. sleep, exercise).
11. Demonstration of proper mental status and cognition for the study
12. Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol
13. If on a non-insulin hyperglycemic therapy, stability on that therapy for the prior 3 months and willingness not to alter the therapy for the study duration.

Exclusion Criteria:

1. Medical need for chronic acetaminophen
2. Use of any medication that at the discretion of the clinical protocol chair is deemed to interfere with the trial.
3. Current treatment of a seizure disorder.
4. Coronary artery disease or heart failure, unless written clearance is received from a cardiologist.
5. Hemophilia or any other bleeding disorder
6. A known medical condition, which in the opinion of the investigator or designee, would put the participant or study at risk such as the following examples:

   1. Inpatient psychiatric treatment in the past 6 months
   2. Presence of a known adrenal disorder
   3. Abnormal liver function test results (Transaminase >3 times the upper limit of normal)
   4. Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2).
   5. Active gastroparesis requiring medical therapy
   6. Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L).
   7. Abuse of alcohol or recreational drugs
   8. Infectious process not anticipated to be resolved prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis, deep tissue infection).
   9. Uncontrolled arterial hypertension (Resting diastolic blood pressure >100 mmHg and/or systolic blood pressure >180 mmHg).
   10. Uncontrolled microvascular complications such as current active proliferative diabetic retinopathy defined as proliferative retinopathy requiring treatment (e.g. laser therapy or VEGF inhibitor injections) in the past 12 months.
7. A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol.
8. Current use of the following drugs and supplements:

   k. Regular acetaminophen user, or not willing to suspend acetaminophen 24 hours before and during the entire length of the trial l. Oral steroids m. Any other medication that the investigator believes is a contraindication to the subject's participation
9. Participation in another pharmaceutical or device trial at the time of enrollment or during the study

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey M. Anderson, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
pending

REFERENCES:
- [Result] Bisio A, Anderson S, Norlander L, O'Malley G, Robic J, Ogyaadu S, Hsu L, Levister C, Ekhlaspour L, Lam DW, Levy C, Buckingham B, Breton MD. Impact of a Novel Diabetes Support System on a Cohort of Individuals With Type 1 Diabetes Treated With Multiple Daily Injections: A Multicenter Randomized Study. Diabetes Care. 2022 Jan 1;45(1):186-193. doi: 10.2337/dc21-0838. PMID 34794973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 111 individuals with T1D on MDI treatment were recruited: 55 at the University of Virginia, 25 at Stanford University, and 31 at the Icahn School of Medicine at Mount Sinai. Across all sites, 12 did not meet the inclusion criteria, and 19 dropped out or withdrew from the trial. The final sample included 80 participants: 23 participants were randomly assigned to the control group (MDI 1 CGM) and 57 to the experimental group (DSS 1 MDI 1 CGM).
Pre-assignment Details: Prior to randomization, the subject initiated a 2 weeks of home use of blinded CGM for characterization of baseline glycemic control and collection of baseline CGM data. The subject used carbohydrate counting per their usual routine with their usual home insulins during this time.
Period: Overall Study
Arm/Group | Continuous Glucose Monitor (CGM)+Decision Support System (DSS) | Continuous Glucose Monitor (CGM) Alone
Started | 57 | 23
Completed | 57 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Monitor (CGM)+Decision Support System (DSS) | Continuous Glucose Monitor (CGM) Alone | Total
Number analyzed (Participants) | 57 | 23 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.44 (14.15) | 39.91 (16.06) | 35.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 11 | 45
  Male | 23 | 12 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 44 | 21 | 65
  African Americans | 5 | 0 | 5
  Asian | 2 | 0 | 2
  Hispanic | 4 | 2 | 6
  Pacific Islander | 1 | 0 | 1
  Alaskan Indian | 1 | 0 | 1
Baseline HbA1c % [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] | 7.41 (1.18) | 7.68 (1.29) | 7.49 (1.21)
Time since T1D diagnosis [Mean (Standard Deviation); unit: years] | 15.85 (12.58) | 15.26 (13.00) | 15.68 (12.62)
Body Mass Index (BMI), kg/m2 [Mean (Standard Deviation); unit: kg/m^2] | 27.42 (5.77) | 26.91 (6.85) | 27.27 (6.06)
Total Daily Insulin, units/kg [Mean (Standard Deviation); unit: units/kg/day] | 0.71 (0.26) | 0.72 (0.30) | .71 (.27)
Continuous Glucose Monitor naive [Count of Participants; unit: Participants] | 27 | 12 | 39
Participants splitting basal insulin into two injections, % [Number; unit: percentage of participants] | 22.9 | 34.8 | 26.3

OUTCOME MEASURES:

1. Primary Outcome: % Time Within Target Range
Description: The primary efficacy outcome is increased % time within target range defined as CGM readings of 70-180 mg/dL.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of time in range
Arm/Group | Continuous Glucose Monitor (CGM)+Decision Support System (DSS) | Continuous Glucose Monitor (CGM) Alone
Number analyzed (Participants) | 57 | 23
percentage of time in range | 57.7 (16.3) | 58.2 (18.8)

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: A reportable adverse event for this protocol includes any untoward medical occurrence that meets criteria for a serious adverse event or any unanticipated medical occurrence in a study subject that is study- or device-related, including severe hypoglycemia and severe hyperglycemia/diabetic ketoacidosis (DKA). Skin reactions from sensor placement are only reportable if severe and/or required treatment.
Arm/Group | Continuous Glucose Monitor (CGM)+Decision Support System (DSS) | Continuous Glucose Monitor (CGM) Alone
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/23
Other Adverse Events (participants affected / at risk) | 0/57 | 0/23

LIMITATIONS AND CAVEATS:
Target enrollment was not reached. Experienced larger-than-expected attrition and, therefore, did not achieve the originally intended statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT03093636/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03093636/ICF_002.pdf